CLINICAL TRIAL: NCT06252818
Title: Validation of a Digital Platform for Functional Respiratory Rehabilitation (ReHub)
Brief Title: Validation of a Digital Platform for Functional Respiratory Rehabilitation
Acronym: ReHub
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bio-Sensing Solutions S.L. (DyCare) (Industry)
Collaborators: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Centre de Validació Clínica de Solucions Digitals (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CVCSD_2301
Record Dates: First submitted 2024-01-24; First posted 2024-02-12 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: ReHub is a medical device designed to assist rehabilitation professionals by providing information for the design, monitoring, and analysis of therapeutic exercise programs for respiratory functional rehabilitation. Patients use the platform to follow the exercise program designed by their therapist from the location that suits them best.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ReHub (Experimental): ReHub is a medical device designed to assist rehabilitation professionals by providing information for the design, monitoring, and analysis of therapeutic exercise programs for respiratory functional rehabilitation. Patients use the platform to follow the exercise program designed by their therapist from the location that suits them best.
  Interventions: Device: ReHub

INTERVENTIONS:
Device: ReHub — ReHub provides support to rehabilitation professionals by offering information for the design, monitoring, and analysis of therapeutic exercise programs for respiratory functional rehabilitation.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD), characterized by persistent airflow limitation in the respiratory airways, is a chronic condition that affects millions of people worldwide. ReHub enables healthcare professionals to design therapeutic exercise programs for the treatment of COPD patients, as well as to analyze and monitor patient rehabilitation through the information and feedback provided via the platform. The main objective of the study is to evaluate the satisfaction and usability of the ReHub platform (for respiratory rehabilitation) among COPD patients and healthcare professionals. This is a single-center satisfaction and usability study on the usage and experience of the ReHub platform (for respiratory rehabilitation).

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD), characterized by persistent airflow limitation in the respiratory airways, is a chronic condition that affects millions of people worldwide. According to various studies, COPD is one of the leading causes of morbidity and mortality in Spain and the third leading cause of death globally. Research conducted in Spain on a representative sample of the population indicates that the overall prevalence of COPD in Spain is approximately 10.2% among adults aged 40 and older. However, significant regional differences are observed, with higher rates in the northern and northeastern regions of the country.

ReHub allows healthcare professionals to design therapeutic exercise programs for the treatment of COPD patients and to analyze and monitor patient rehabilitation through the information and feedback provided via the platform.

The main objective of the study is to assess the satisfaction and usability of the ReHub platform (for respiratory rehabilitation) among COPD patients and healthcare professionals.

Methology:

Single-center satisfaction and usability study on the usage and experience of the ReHub platform (for respiratory rehabilitation). Additionally, changes in clinical parameters and functional status will be evaluated at the end of the study compared to the baseline situation (pre-post intervention study without a control group).

Recruitment will take place at the Respiratory Rehabilitation Service of Hospital Sant Pau (Barcelona-Spain). A consecutive sampling of patients who meet the inclusion criteria will be conducted during the recruitment period or until the sample size of 100 participants is reached. Participants who meet the inclusion criteria and none of the exclusion criteria will be invited to participate in the study. Once their acceptance to participate is obtained, they will be included in the study and will receive training on how to use the ReHub platform.

After using the platform for a minimum of 4 months, a survey will be administered to the patients to assess their satisfaction and usability. Additionally, changes in clinical parameters and the functional status of the patients will be assessed at the end of the study compared to the baseline situation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD, GOLD grade I - IV
* Need of respiratory rehabilitation.
* 18 years of age or older.
* Explicit willingness to participate in the study.
* Diagnosis of COPD (FEV1/FVC < 70)

Exclusion Criteria:

* Individuals with cognitive impairment.
* Language barriers or illiteracy (inability to read in Spanish).
* Lack of access to a mobile device with an internet connection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale (SUS) | 4 months
  User satisfaction and experience (Spanish version), from 0 to 100; higher score means a better outcome
Satisfaction and Usability Questionnaire with Comprehensive Outpatient follow-up health applications (pSUAPP-S) for Patients | 4 months
  Satisfaction and Usability Questionnaire with Comprehensive Outpatient follow-up health applications for patients, from 0 to 100; higher score means a better outcome
Satisfaction and Usability Questionnaire with Comprehensive Outpatient follow-up health applications (pSUAPP-S) for Healthcare Professionals | 4 months
  Satisfaction and Usability Questionnaire with Comprehensive Outpatient follow-up health applications for Healthcare professionals, from 0 to 100; higher score means a better outcome

SECONDARY OUTCOMES:
Walking test_dysnea | Baseline and 4 months
  Dyspnea level (pre and post) assessed by Borg Scale (number from 0 none to 10 maximum)
Walking test_fatigue | Baseline and 4 months
  Fatigue level (pre and post) assessed by Borg Scale (number from 0 none to 10 maximum)
Walking test_oxygen | Baseline and 4 months
  SaO2 (oxygen saturation) (pre and post) in percent
Walking test_ heart rate | Baseline and 4 months
  Heart rate (pre and post) in beats per minute (bpm)
Walking test_distance | Baseline and 4 months
  Distance walked in meters
Walking test_stops | Baseline and 4 months
  Number of stops (integer number)
Walking test_stops duration | Baseline and 4 months
  Stops duration in minutes
Adverse events during exercise | During the exercises
  Adverse events during exercise: dyspnea (shortness of breath)
Adherence to the platform_frequency | 4 months
  Compliance with the rehabilitation program in terms of frequency of use (number of days connected to the platform)
Adherence to the platform_compliance | 4 months
  Compliance with the rehabilitation program in terms of percent of performed exercices versus prescribed exercices
Adherence to the platform_connection time | 4 months
  Compliance with the rehabilitation program in terms of connection time (in minutes)
Interaction between the physiotherapist and the patient | During the follow-up until 4 months
  Number of messages exchanged between the patient and the physiotherapist through ReHub platform
Chronic Obstructive Pulmonary Disease (COPD) Assessment scale (CAT) | Baseline and 4 months
  Quality of life COPD patients scale; from 0 to 40; higher score means a worse outcome
modified Medical Research Council scale (mMRC) | Baseline and 4 months
  Dyspnea scale; from 0 to 4; higher score means a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Carme Puy, MD, Principal Investigator — Pneumologist at Hospital Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No